CLINICAL TRIAL: NCT05530161
Title: Effect of Hypocalcemia on the Outcome of Elderly Major Trauma Patients With Trauma-induced Coagulopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-822
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Coagulopathy; Trauma
Keywords: trauma
MeSH Terms: conditions — Hemostatic Disorders; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- trauma induced coagulopathy: patients with INR>1.2
  Interventions: Other: hypocalcemia
- non-trauma induced coagulopathy: patients with INR≤1.2

INTERVENTIONS:
Other: hypocalcemia — hypocalcemia or normocalcemia
  Groups: trauma induced coagulopathy

SUMMARY:
Hypocalcaemia is an independent risk factor of TIC in elderly trauma patients. TIC combined with hypocalcemia had worse coagulation function and more serious acidosis.

DETAILED DESCRIPTION:
This 5-year retrospective, observational, single-center study was conducted at the Second Affiliated Hospital of Zhejiang University Medical School (SAHZU, China). Elderly patients with trauma were registered when they were admitted into intensive care unit affiliated to department of Emergency medicine (EICU) since January 2015 and September 2020.The purpose of this study is to elucidate the effect of hypocalcemia on TIC in elderly trauma patients through a single-center retrospective study, so as to further optimize the diagnosis and treatment strategies for TIC in elderly trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* age≥65 years old
* history of trauma

Exclusion Criteria:

* previous anticoagulants or antiplatelet medication;
* Coagulopathy caused by previous underlying diseases;
* Blood products transfused before admission;
* Cardiac arrest on admission;
* Malignant tumor;
* Data incomplete

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with trauma were registered when they were admitted into intensive care unit affiliated to department of Emergency medicine (EICU) since January 2015 and September 2020
Sampling Method: Probability Sample
Enrollment: 371 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Internationalized Normalized Ratio (INR) | 24 hour
  coagulation function :Internationalized Normalized Ratio (INR)
Activated Partial Thromboplastin Time (APTT) | 24 hour
  coagulation function : Activated Partial Thromboplastin Time (APTT)
Prothrombin Time (PT) | 24 hour
  coagulation function : Prothrombin Time (PT)

SECONDARY OUTCOMES:
Blood products rate | through study completion, an average of 1 week
  the rate of Blood products use

CONTACTS AND LOCATIONS:
Overall Officials: yongan xu, doctor, Study Chair — Department of Emergency medicine，Second Affiliated Hospitalof Zhejiang University
Locations (1):
- SAHZU, Hanzhou, Zhejiang, China